CLINICAL TRIAL: NCT01239121
Title: Implementing a Regional Data Exchange Tool to Improve Medication Use and Safety
Brief Title: Regional Data Exchange to Improve Medication Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Victoria (Other); Weill Medical College of Cornell University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 10-146
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Drug Toxicity
Keywords: drug toxicity; drug interactions; electronic health records; medical errors
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HIE-Enhanced Medication Reconciliation (Experimental): Health Information Exchange (HIE)-Enhanced Medication Reconciliation for Veterans admitted to James J Peters VA hospital units 6B, 7B, 7C, and 8B (each unit crossing over between intervention and control every 3-4 months)
  Interventions: Other: HIE-Enhanced Medication Reconciliation
- Optimal Medication Reconciliation without HIE (Active Comparator): Optimal Medication Reconciliation without Health Information Exchange (HIE) for Veterans admitted to James J Peters VA hospital units 6B, 7B, 7C, and 8B (each unit crossing over between intervention and control every 3-4 months)
  Interventions: Other: Optimal Medication Reconciliation without HIE
- Pilot HIE-Enhanced Outpatient Medication Reconciliation (Other): Health Information Exchange (HIE)-Enhanced Medication Reconciliation for Veterans seen as outpatients in Geriatrics Primary care clinic
  Interventions: Other: HIE-Enhanced Medication Reconciliation

INTERVENTIONS:
Other: HIE-Enhanced Medication Reconciliation — Medication reconciliation enhanced by regional health information exchange, implemented by a pharmacist
  Arms: HIE-Enhanced Medication Reconciliation; Pilot HIE-Enhanced Outpatient Medication Reconciliation
Other: Optimal Medication Reconciliation without HIE — Medication reconciliation implemented by a pharmacist without regional health information exchange
  Arms: Optimal Medication Reconciliation without HIE

SUMMARY:
Medication reconciliation, a process by which a provider obtains and documents a thorough medication history with specific attention to comparing current and previous medication use, can prevent medication-related errors and harm. The aims of this study are: 1) To adapt medication reconciliation to include information from a computerized regional health information exchange (RHIO) in the Bronx, 2) To conduct a trial of the adapted medication reconciliation process and examine effects on medication errors, harm, and hospital costs, and 3) To identify factors that are barriers to adoption of the RHIO tool by James J. Peters (Bronx) VA providers. Findings from this project will provide an understanding of the effect of the RHIO tool on reducing harmful VA and non-VA medication use. It will also provide information on the feasibility of incorporating RHIO tool use into every day work flow for pharmacists and physicians.

DETAILED DESCRIPTION:
Medication reconciliation, a process by which a provider obtains and documents a thorough medication history with specific attention to comparing current and previous medication use, can prevent medication-related errors and harm. The most important barrier to effective medication reconciliation is the unreliability of patients' own reports about their medication use and incomplete provider history-taking. The James J. Peters VA (JJP VA) participates in the Bronx RHIO, a New York State-funded health information exchange organization that in October 2008 implemented clinical data information exchange among the largest healthcare providers in the Bronx. JJP VA providers can now access clinical data, including medication use, from non-VA facilities with patients' consent. The aims of this study are: 1) To adapt a medication reconciliation process to include information from a regional health information exchange (RHIO), 2) To conduct a controlled trial of a medication reconciliation process at the time of hospital admission either enhanced or not enhanced with data from a regional health information exchange, and examine effects on transition drug risk, adverse drug events, and total inpatient costs, and 3) To identify system and provider factors that impede and facilitate adoption of the information exchange tool for routine use by VA providers. The investigators plan to conduct qualitative and quantitative studies. First the investigators will perform cognitive task analysis (CTA) to examine providers' decision-making and to map RHIO tool functions while providers interface with the tool, with interview questions to identify factors that facilitate or hinder use. Second, the investigators will enroll patients admitted to 2 inpatient units at the JJP VA, and assign them to receive usual medication reconciliation or RHIO-enhanced medication reconciliation with a notification to physicians about the patient's non-VA services that can be viewed in the RHIO. The investigators will measure transition drug risk and ADEs by medical record review and patient interview, and measure inpatient costs with administrative cost data from national VA datasets. Third, the investigators will conduct CTA with pharmacists and physicians at the end of the quantitative study who are expert in use of the tool to characterize differences in cognitive processes from prior to the quantitative study. This will supply information on system and provider factors that impede and facilitate adoption of the tool for routine use, and on potential improvements in the tool. Findings from this project will provide an understanding of the effect of real-time review of Veteran's non-VA medication use -- enabled by a Regional Health Information Organization (RHIO) tool -- on reducing duplicative VA and non-VA medication use and adverse drug events in Veterans. It will also provide information on the feasibility and effectiveness of incorporating RHIO tool access and use into every day work flow for VA pharmacist and physician providers.

ELIGIBILITY:
Inclusion Criteria:

* Veterans admitted to James J. Peters VA hospital units 6B, 7B, 7C, or 8B or seen as outpatients in the Geriatrics Primary care clinic, who have an identity match in the Bronx RHIO, who consent to participate in the Bronx RHIO, and who stay on the unit at least 24 hours

Exclusion Criteria:

* Cannot be transferred from another James J. Peters VA hospital unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Boockvar, MD MS, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung WW, Morano B, Moodhe N, Boockvar K. Regional Health Information Organization (RHIO): its potential uses to improve veteran health care. Federal practitioner : for the health care professionals of the VA, DoD, and PHS. 2011 Jan 1; 28(3):33-36.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIE-Enhanced Medication Reconciliation | Optimal Medication Reconciliation Without HIE | Pilot HIE-Enhanced Outpatient Medication Reconciliation
Started | 188 | 199 | 15
Completed | 186 | 195 | 15
Not Completed | 2 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIE-Enhanced Medication Reconciliation | Optimal Medication Reconciliation Without HIE | Pilot HIE-Enhanced Outpatient Medication Reconciliation | Total
Number analyzed (Participants) | 186 | 195 | 15 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (14.4) | 60.8 (14.5) | 86.4 (6.8) | 60.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 0 | 13
  Male | 180 | 188 | 15 | 383
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 55 | 1 | 100
  Not Hispanic or Latino | 138 | 138 | 11 | 287
  Unknown or Not Reported | 4 | 2 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 1 | 4
  Black or African American | 121 | 120 | 4 | 245
  White | 57 | 64 | 9 | 130
  More than one race | 1 | 3 | 1 | 5
  Unknown or Not Reported | 6 | 6 | 0 | 12
Region of Enrollment [Number; unit: participants]
  United States | 186 | 195 | 15 | 396

OUTCOME MEASURES:

1. Primary Outcome: Transition Drug Risk
Description: Rating of potential for harm to patient from hospital medication discrepancies by record review. Minimum=0 Maximum=no maximum. Higher values represent increased detection of medication discrepancies. Although medication discrepancies are undesirable, increasing their detection might facilitate prevention of adverse drug events.
Time Frame: During hospital stay and up to 1 month after hospital discharge
Population: Outcome not ascertained in the third arm because those participants were not hospitalized.
Measure: Mean (Standard Deviation); unit: units: risk-weighted discrepancies
Arm/Group | HIE-Enhanced Medication Reconciliation | Optimal Medication Reconciliation Without HIE | Pilot HIE-Enhanced Outpatient Medication Reconciliation
Number analyzed (Participants) | 186 | 195 | 0
units: risk-weighted discrepancies | 6.4 (5.9) | 5.8 (5.0) |
Statistical Analysis 1: Comparison: HIE-Enhanced Medication Reconciliation vs Optimal Medication Reconciliation Without HIE; Test type: Superiority or Other; p = 0.175, Regression, Linear; Slope = 0.60, 95% CI 2-sided [-0.27 to 1.5]

2. Secondary Outcome: Adverse Drug Events
Description: Actual harm to patient from hospital medication discrepancies by record review
Time Frame: During hospital stay and up to 1 month after hospital discharge
Population: Outcome not ascertained in the third arm because those participants were not hospitalized.
Measure: Number; unit: participants
Arm/Group | HIE-Enhanced Medication Reconciliation | Optimal Medication Reconciliation Without HIE | Pilot HIE-Enhanced Outpatient Medication Reconciliation
Number analyzed (Participants) | 186 | 195 | 0
participants | 19 | 18 |
Statistical Analysis 1: Comparison: HIE-Enhanced Medication Reconciliation vs Optimal Medication Reconciliation Without HIE; Test type: Superiority or Other; p = 0.964, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [.49 to 2.1]

3. Secondary Outcome: Medication-related Symptoms
Description: Patient's self-report of medication-related symptoms by telephone questionnaire
Time Frame: Up to 1 month after hospital discharge
Population: For this outcome 66 and 87 participants unable to be reached by telephone in first and second arms, respectively.
  Outcome not ascertained in the third arm because those participants were not hospitalized.
Measure: Number; unit: participants
Arm/Group | HIE-Enhanced Medication Reconciliation | Optimal Medication Reconciliation Without HIE | Pilot HIE-Enhanced Outpatient Medication Reconciliation
Number analyzed (Participants) | 120 | 108 | 0
participants | 24 | 21 |

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events during the hospital stay (up to a maximum of 30 days) and up to 30 days after hospital discharge.
Arm/Group | HIE-Enhanced Medication Reconciliation | Optimal Medication Reconciliation Without HIE | Pilot HIE-Enhanced Outpatient Medication Reconciliation
Serious Adverse Events (participants affected / at risk) | 39/186 | 36/195 | 0/15
Other Adverse Events (participants affected / at risk) | 24/120 | 21/108 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIE-Enhanced Medication Reconciliation (N=186) | Optimal Medication Reconciliation Without HIE (N=195) | Pilot HIE-Enhanced Outpatient Medication Reconciliation (N=15)
Hospital Readmission (Investigations) | 39 | 36 | 0 — Outcome not ascertained in the third arm because those participants were not hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIE-Enhanced Medication Reconciliation (N=120) | Optimal Medication Reconciliation Without HIE (N=108) | Pilot HIE-Enhanced Outpatient Medication Reconciliation (N=0)
Medication-related symptoms (Investigations) | 24 | 21 | 0 — For this outcome 66 and 87 participants unable to be reached by telephone in first and second arms, respectively.Outcome not ascertained in the third arm because those participants were not hospitalized.

LIMITATIONS AND CAVEATS:
In the HIE-enhanced medication reconciliation intervention arm, the Health Information Exchange (HIE) capabilities were reduced from what was planned, limiting the potency of the intervention relative to control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes